CLINICAL TRIAL: NCT02724774
Title: Collaborative Perinatal Mental Health and Parenting Support in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susan Spieker, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00010114; R01HD080851 (NIH)
Record Dates: First submitted 2016-03-15; First posted 2016-03-31 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Parenting; Mother-child Relations
Keywords: infants; mental health; postpartum period
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promoting First Relationships® (PFR) (Experimental): 10 week home visiting program
  Interventions: Behavioral: Promoting First Relationships®
- Parent Information Packet (No Intervention): A packet is mailed to the families, including handouts related to child development, health, and local resources.

INTERVENTIONS:
Behavioral: Promoting First Relationships® — PFR is based on attachment theory and is strengths-based. The 10 week intervention is delivered in the home of the family. Each week has a theme for discussion, handouts, an activity, and time for "joining" - checking in with the parent, listening to her concerns, and establishing a positive, supportive relationship. The PFR provider videotapes playtime between parent and child, and alternates every other week with watching the video with the parent, reflecting about the needs of both parent and child. The provider helps the parent develop greater empathy and understanding of the child's needs and feelings, and helps the parent to identify her own feelings and needs around parenting.
  Other Names: PFR
  Arms: Promoting First Relationships® (PFR)

SUMMARY:
Treating mothers' perinatal depressive and other mental health symptoms alone does not prevent impaired parenting quality and adverse infant outcomes. The goal of this research is to conduct a randomized controlled trial to evaluate the effectiveness of adding a research-based 10-week home visiting parenting program to evidence-based mental health treatment, to counter the pernicious effects of mothers' symptoms on parenting quality and infant development. Participants will be English and Spanish-speaking low-income mothers who began publicly funded mental/behavioral health treatment in pregnancy at their primary care community health centers.

DETAILED DESCRIPTION:
Infants exposed to impaired parenting as a result of their mothers' major depression and other mental health disorders in the perinatal period are at risk for compromised social interaction and affective and behavioral regulation. Depression is the most frequently reported mental health condition during the perinatal period; about 9% of infants under one year have mothers who experience a major depressive episode. That rate nearly triples to 25% for infants of mothers below 200% of the federal poverty level. In addition to poverty, young maternal age, lack of social support, low education, and adverse childhood experiences are all risk factors for depression, anxiety, and other mental health conditions. Two strands of research point to the need for effective parenting support for mothers following treatment for mental health conditions in pregnancy. First, depressed mothers frequently fail to accurately notice, interpret, or respond sensitively to infant cues. Alarmingly, mothers' impaired parenting of their infants continues even after their depression has been successfully treated. Second, newborns of prenatally depressed women are physiologically dysregulated and hence more challenging to nurture. With the passage of the Affordable Care Act and Maternal, Infant, and Early Childhood Home Visiting, the federal government is supporting states to implement high-quality home visiting programs as part of a comprehensive early childhood system for vulnerable families experiencing the risk factors associated with maternal depression and other mental health symptoms. But two important limitations of home visiting have been identified: child development home visitors are not trained to deal meaningfully with maternal depression and other mental health conditions, and they are often not sufficiently trained to support infant-mother relationships. Our study has the potential to inform intervention programs nationwide by testing the effectiveness of adding a short, attachment-based, home-visiting parenting program to an existing, evidence-based mental health treatment program delivered via community primary care clinics serving pregnant and parenting women from vulnerable populations. The goal of this research is to conduct a randomized controlled trial to evaluate the effectiveness of Promoting First Relationships® for English and Spanish-speaking low-income mothers who were treated for depression or other mental health conditions beginning in pregnancy and as needed in the perinatal year. Treatment will be coordinated through the publicly funded, evidenced-based Mental Health Integration Program for High-Risk Pregnant and Parenting Women (MHIP Moms) in primary care community health centers that target safety-net populations in King County, Washington. Promoting First Relationships® is a research-based, 10-week home visiting program that uses video feedback and strengths-based consultation strategies to increase mothers' parenting competence and confidence. Bilingual community providers will deliver Promoting First Relationships® after a baseline assessment and random assignment at infant age three months. Post tests will occur at infant age six and twelve months. The primary specific aims are to test the effectiveness of PFR to improve parenting quality for low income, English and Spanish speaking mothers who began mental/behavioral health treatment during pregnancy, and to improve social and regulatory outcomes for their infants.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with infants 6 weeks - 3 months old
* English or Spanish speaking
* Access to a telephone
* Currently or at some point during pregnancy received treatment for a mental health condition (counseling and/or medications) at a participating community health center in the Seattle, Washington area

Exclusion Criteria:

* Currently experiencing an acute crisis (e.g., severe domestic violence, homelessness, hospitalization, imprisonment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Spieker, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnard, K. E. (1994). What the Teaching Scale measures. In G. S. Sumner & A. Spietz (Eds.), NCAST: Caregiver/parent-child interaction teaching manual. University of Washington NCAST Publications.
- [Background] Kelly, J., & Korfmacher, J. (2008). Raising a baby. University of Washington NCAST Publications.
- [Background] Kelly, J., Sandoval, D., Zuckerman, T. G., & Buehlman, K. (2008). Promoting First Relationships: A program for service providers to help parents and other caregivers nurture young children's social and emotional development (2 ed.). University of Washington NCAST Programs.
- [Background] Zahr LK. The relationship between maternal confidence and mother-infant behaviors in premature infants. Res Nurs Health. 1991 Aug;14(4):279-86. doi: 10.1002/nur.4770140406. PMID 1891613
- [Background] Crittenden, P. M. (1979-2010). CARE-Index: Infant Coding Manual. Family Relations Institute.
- [Background] Carter AS, Briggs-Gowan MJ, Jones SM, Little TD. The Infant-Toddler Social and Emotional Assessment (ITSEA): factor structure, reliability, and validity. J Abnorm Child Psychol. 2003 Oct;31(5):495-514. doi: 10.1023/a:1025449031360. PMID 14561058
- [Result] Oxford ML, Hash JB, Lohr MJ, Bleil ME, Fleming CB, Unutzer J, Spieker SJ. Randomized trial of promoting first relationships for new mothers who received community mental health services in pregnancy. Dev Psychol. 2021 Aug;57(8):1228-1241. doi: 10.1037/dev0001219. PMID 34591567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in collaboration with the Mental Health Integration Program (MHIP) and Maternity Support Services (MSS) of Public Health Seattle and King County, Washington. Five community health clinics offering MHIP agreed to assist in study recruitment. Eligible participants received mental health treatment during pregnancy, spoke English or Spanish, had an infant under three months, had a telephone, and were planning to remain in the study area until the child's first birthday.
Pre-assignment Details: 599 cases were screened for eligibility. 353 were determined eligible and contacted about the study 101 declined (74 not interested; 20 unreachable; 7 could not be enrolled because at that time there was no space in the program). 252 were seen in the baseline visit and randomized.
Period: Overall Study
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Started | 127 | 125
Infant 6 Months | 122 | 122
Infant 12 Months | 120 | 123
Completed | 120 | 123
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Population: Mother-infant dyads were recruited and randomized in pairs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet | Total
Number analyzed (Participants) | 127 | 125 | 252
Age, Categorical [Count of Participants; unit: Participants] — Population: Each arm consisted of dyads of mother-infant pairs.
  Participants
    Mothers: <=18 years | 0 | 0 | 0
    Mothers: Between 18 and 65 years | 127 | 125 | 252
    Mothers: >=65 years | 0 | 0 | 0
    Infants: <=18 years | 127 | 125 | 252
    Infants: Between 18 and 65 years | 0 | 0 | 0
    Infants: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Mother's age is in years. Population: The full sample consists of 252 mothers and 252 infants, or 504 individuals. Mother-infant dyads were randomized in pairs, 127 to PFR, 125 to the control arm.
  years
    Mother participants | 28.8 (5.8) | 27.4 (5.6) | 28.07 (5.8)
    Infant participants | .15 (.04) | .15 (.04) | .15 (.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 504 study participants consisting of 252 mother-infant dyads.
  Participants
    Sex: Mothers: Female | 127 | 125 | 252
    Sex: Mothers: Male | 0 | 0 | 0
    Sex: Infants: Female | 56 | 64 | 120
    Sex: Infants: Male | 71 | 61 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  mothers: Hispanic or Latino | 62 | 57 | 119
  mothers: Not Hispanic or Latino | 65 | 68 | 133
  mothers: Unknown or Not Reported | 0 | 0 | 0
  infants: Hispanic or Latino | 68 | 66 | 134
  infants: Not Hispanic or Latino | 59 | 59 | 118
  infants: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Mothers: American Indian or Alaska Native | 2 | 2 | 4
  Mothers: Asian | 3 | 5 | 8
  Mothers: Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Mothers: Black or African American | 21 | 23 | 44
  Mothers: White | 84 | 81 | 165
  Mothers: More than one race | 16 | 10 | 26
  Mothers: Unknown or Not Reported | 0 | 1 | 1
  Infants: American Indian or Alaska Native | 1 | 4 | 5
  Infants: Asian | 2 | 0 | 2
  Infants: Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Infants: Black or African American | 20 | 17 | 37
  Infants: White | 79 | 68 | 147
  Infants: More than one race | 25 | 33 | 58
  Infants: Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Data are reported in dyads consisting of mother-infant pairs
  participants
    United States | 127 | 125 | 252
NCATS Parenting Sensitivity [Mean (Standard Deviation); unit: units on a scale] — Nursing Child Assessment Teaching Scale: coded from observation of mother interacting with infant during teaching task (NCATS; Barnard, 1994). The parenting sensitivity score can range from 0 to 50; higher scores indicate greater sensitivity. Population: Missing data
  units on a scale
    number analyzed (Participants) | 125 | 123 | 248
    (all) | 35.13 (4.90) | 34.21 (5.13) | 34.63 (4.97)
Sensitivity in Play-Dyadic Synchrony [Mean (Standard Deviation); unit: units on a scale] — Child-Adult Relationship Experimental-Index (CARE-Index): coded from observation of mother and infant in free play activity (Crittenden, 1979-2005). Dyadic synchrony and maternal sensitivity scores can range from 0 to 14, with higher scores indicating more positive interactions. [Because maternal sensitivity and dyadic synchrony are correlated .98-.99, only dyadic synchrony will be reported.] Population: Missing data
  units on a scale
    number analyzed (Participants) | 126 | 125 | 251
    (all) | 4.58 (2.41) | 3.88 (2.13) | 4.26 (2.32)
Parent Understanding of Toddlers [Mean (Standard Deviation); unit: units on a scale] — Raising a Baby Scale (Kelly, Korfmacher, & Buehlman, 2008): 16-item self report measure rated on a 4-point agree/disagree scale. The scores can range from 16 to 64, with higher scores indicating greater parental knowledge. Population: Missing data
  units on a scale
    number analyzed (Participants) | 127 | 124 | 251
    (all) | 51.17 (5.05) | 49.88 (4.98) | 50.66 (5.18)
Maternal Confidence [Mean (Standard Deviation); unit: units on a scale] — Maternal Confidence Questionnaire (MCQ; Zahr, 1991): 14-item self report measure rated on a 5-point frequency scale. The mean score can range from 1 to 5, with higher scores indicating greater maternal confidence.
  units on a scale | 4.23 (.44) | 4.19 (.48) | 4.21 (.46)
Infant Interactive Quality-Difficultness [Mean (Standard Deviation); unit: units on a scale] — CARE-Index: coded from observation of mother and infant in free play activity (Crittenden, 1979-2005). Child cooperation scores can range from 0 to 14, with higher scores indicating more positive interactions. (Because child cooperation and dyadic synchrony are correlated .95-.96, a different CARE-Index scale with lower correlations with dyadic synchrony (-.32 to .05), child difficultness, will be used). Population: Missing data
  units on a scale
    number analyzed (Participants) | 126 | 125 | 251
    (all) | 3.81 (3.26) | 4.12 (3.03) | 4.02 (3.13)

OUTCOME MEASURES:

1. Primary Outcome: Change in Parent Sensitivity in Teaching
Description: Nursing Child Assessment Teaching Scale: coded from observation of mother interacting with the infant during teaching task. The parenting sensitivity score can range from 0 to 50; higher scores indicate greater sensitivity.
Time Frame: Baseline to infant age 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 113 | 112
score on a scale | 36.73 (4.30) | 35.32 (4.52)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; All analyses were conducted as intention-to-treat, analyzing all 252 cases as randomly assigned to the PFR and control group (CG). Multiple linear regression was used to examine the treatment effect of PFR (0 = CG, 1 = PFR). Covariates included preferred language (0 = English, 1 = Spanish) and the baseline measure; Test type: Superiority; p = .026, Regression, Linear — a priori threshold for statistical significance p < .05

2. Primary Outcome: Change in Parent Sensitivity in Play
Description: Child-Adult Relationship Experimental-Index (CARE-Index): coded from observation of mother and infant in free play activity. Dyadic synchrony and maternal sensitivity scores can range from 0 to 14, with higher scores indicating more positive interactions. [Because maternal sensitivity and dyadic synchrony are correlated .98-.99, only dyadic synchrony will be reported.]
Time Frame: Baseline to infant age 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 113 | 112
units on a scale | 6.45 (2.12) | 5.98 (2.35)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; Test type: Superiority; p = .154, Regression, Linear — a priori threshold for statistical significance p < .05

3. Primary Outcome: Change in Maternal Confidence
Description: Maternal Confidence Questionnaire (MCQ; Zahr, 1991): 14-item self report measure rated on a 5-point frequency scale. The mean score can range from 1 to 5, with higher scores indicating greater maternal confidence.
Time Frame: Baseline to infant age 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 120 | 123
score on a scale | 4.40 (.33) | 4.36 (.37)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; Test type: Superiority; p = .516, Regression, Linear — a priori threshold for statistical significance p < .05

4. Primary Outcome: Change in Parent Understanding of Toddlers
Description: Raising a Baby Scale: 16-item self-report measure rated on a 4-point agree/disagree scale. The scores can range from 16 to 64, with higher scores indicating greater parental knowledge.
Time Frame: Baseline to infant age 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 120 | 123
score on a scale | 51.84 (4.88) | 48.67 (5.06)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; Test type: Superiority; p < 0.001, Regression, Linear — a priori threshold for statistical significance p < .05

5. Secondary Outcome: Change in Infant Interactive Quality
Description: CARE-Index: coded from observation of mother and infant in free play activity. Child cooperation scores can range from 0 to 14, with higher scores indicating more positive interactions. (Because child cooperation and dyadic synchrony are correlated .95-.96, a different CARE-Index scale with lower correlations with dyadic synchrony (-.32 to .05), child difficultness, will be used).
Time Frame: Baseline to infant age 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 113 | 112
units on a scale | 2.23 (2.02) | 2.71 (2.37)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; Test type: Superiority; p = 0.094, Regression, Linear — a priori threshold for statistical significance p < .05

6. Secondary Outcome: Infant Behavioral Regulation: Externalizing T Score
Description: Infant Toddler Social Emotional Assessment: maternal report of child internalizing, externalizing, and dysregulation problem behaviors. T scores can range from 20 to 99, with higher scores indicating more behavior problems.
Time Frame: infant age 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 120 | 123
score on a scale | 59.24 (11.06) | 62.54 (12.37)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; Test type: Superiority; p = 0.029, Regression, Linear

7. Secondary Outcome: Infant Behavioral Regulation: Internalizing T Score
Description: as for outcome 6
Time Frame: infant age 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 120 | 123
score on a scale | 53.64 (10.82) | 54.93 (11.48)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; Test type: Superiority; p = .389, Regression, Linear — a priori threshold for statistical significance p < .05

8. Secondary Outcome: Infant Behavioral Regulation: Dysregulation T Score
Description: as for outcome 6
Time Frame: infant age 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
Number analyzed (Participants) | 120 | 123
score on a scale | 54.82 (13.62) | 55.33 (13.66)
Statistical Analysis 1: Comparison: Promoting First Relationships® (PFR) vs Parent Information Packet; Test type: Superiority; p = .747, Regression, Linear — a priori threshold for statistical significance p < .05

ADVERSE EVENTS:
Time Frame: 12 months
Description: Both groups received positive services and no physical/medical intervention.
Arm/Group | Promoting First Relationships® (PFR) | Parent Information Packet
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/125
Other Adverse Events (participants affected / at risk) | 0/127 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02724774/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02724774/SAP_002.pdf
  • Informed Consent Form (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT02724774/ICF_003.pdf